CLINICAL TRIAL: NCT06673524
Title: Effect of Transversus Abdominis Plan Block and Recto-Intercostal Fascial Plan Block in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Güvenç Doğan, Associate Professor, Hitit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-103
Record Dates: First submitted 2024-11-02; First posted 2024-11-05 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Pain
Keywords: Cholecystectomy; Pain; Postoperative; Transversus Abdominis Plan Block; Recto-Intercostal Fascial Plan Block
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Sensitivity Training Groups

STUDY DESIGN:
Intervention Model Description: TAP Block: Aseptic conditions are established. With the patient supine, the ultrasound (USG) probe is placed laterally to the xiphoid process at the rib cage's lower border, visualizing the rectus abdominis above the transversus abdominis. The internal oblique aponeurosis is seen between the transversus and external oblique muscles. Pressure is applied to optimize myofascial plane visualization. A 22-25G, 50-100 mm block needle is used in an in-plane technique to inject 20 ml of 0.25% bupivacaine in the fascial plane between the rectus and transversus abdominis, then repeated on the opposite side.
  Rectus-Intercostal Fascial Plane Block: With the patient supine under USG, a probe is placed 2-3 cm lateral to the xiphoid process to visualize the rectus abdominis and 6th-7th costal cartilages. A needle is advanced to inject 20 ml of 0.25% bupivacaine into the interfascial plane, repeated on the opposite side.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group T (Transversus Abmoninis Plane Block) (Active Comparator): TAP Block: Aseptic conditions are ensured in the area where the block will be performed. With the patient in the supine position, the ultrasound (USG) probe is placed in an oblique position lateral to the xiphoid process at the lower border of the rib cage. The rectus abdominis muscle and its posterior sheath are visualized above the transversus abdominis muscle. At this level, only the aponeurosis of the internal oblique muscle can be seen between the transversus and external oblique muscles. By applying some pressure and tilt to the probe, the image of the myofascial planes is better optimized. Using a 22-25G, 50-100 mm block needle, an in-plane technique is applied, advancing either medially to laterally or vice versa. In the fascial plane between the rectus abdominis and transversus abdominis or between the internal oblique and transversus abdominis muscles, 20 ml of 0.25% bupivacaine is injected. The same procedure is then applied to the opposite side.
  Interventions: Procedure: Group T (Transversus Abmoninis Plane Block)
- Group R (Rectus-Intercostal Fascial Plane Block) (Active Comparator): Rectus-Intercostal Fascial Plane Block: Aseptic conditions are ensured in the area where the block will be performed. With the patient in the supine position and under ultrasound (USG) guidance, a linear probe is placed 2-3 cm lateral and caudal to the xiphoid process to visualize the rectus abdominis muscle and the 6th-7th costal cartilages. Using an in-plane technique, the needle is advanced from caudal to cephalad. After confirming the target by hydrodissecting between the ribs and the rectus abdominis muscle, 20 ml of 0.25% bupivacaine is injected into the interfascial plane between the 6th-7th ribs and the rectus abdominis muscle using a 22-G, 80 mm block needle. The same procedure is then applied to the opposite side.
  Interventions: Procedure: Group R (Rectus-Intercostal Fascial Plane Block)

INTERVENTIONS:
Procedure: Group T (Transversus Abmoninis Plane Block) — TAP Block: Aseptic conditions are ensured in the area where the block will be performed. With the patient in the supine position, the ultrasound (USG) probe is placed in an oblique position lateral to the xiphoid process at the lower border of the rib cage. The rectus abdominis muscle and its posterior sheath are visualized above the transversus abdominis muscle. At this level, only the aponeurosis of the internal oblique muscle can be seen between the transversus and external oblique muscles. By applying some pressure and tilt to the probe, the image of the myofascial planes is better optimized. Using a 22-25G, 50-100 mm block needle, an in-plane technique is applied, advancing either medially to laterally or vice versa. In the fascial plane between the rectus abdominis and transversus abdominis or between the internal oblique and transversus abdominis muscles, 20 ml of 0.25% bupivacaine is injected. The same procedure is then applied to the opposite side.
  Arms: Group T (Transversus Abmoninis Plane Block)
Procedure: Group R (Rectus-Intercostal Fascial Plane Block) — Rectus-Intercostal Fascial Plane Block: Aseptic conditions are ensured in the area where the block will be performed. With the patient in the supine position and under ultrasound (USG) guidance, a linear probe is placed 2-3 cm lateral and caudal to the xiphoid process to visualize the rectus abdominis muscle and the 6th-7th costal cartilages. Using an in-plane technique, the needle is advanced from caudal to cephalad. After confirming the target by hydrodissecting between the ribs and the rectus abdominis muscle, 20 ml of 0.25% bupivacaine is injected into the interfascial plane between the 6th-7th ribs and the rectus abdominis muscle using a 22-G, 80 mm block needle. The same procedure is then applied to the opposite side.
  Arms: Group R (Rectus-Intercostal Fascial Plane Block)

SUMMARY:
Cholecystectomy is a common surgical procedure performed globally for acute cholecystitis. Management of acute cholecystitis is divided into medical and surgical approaches. Medical management involves bed rest, analgesic agents, antibiotic therapy, and IV fluid replacement. Surgical management includes cholecystectomy, the removal of the gallbladder, which can be done via open surgery or laparoscopically. The laparoscopic approach has advantages over open surgery, such as reduced pain at incision sites, shorter hospital stays, improved quality of life, and faster recovery. However, despite its minimally invasive nature, laparoscopic cholecystectomy (LC) can still cause moderate to severe pain. Severe pain may delay ambulation, reduce patient satisfaction, lead to chronic pain, and increase the risk of pulmonary and cardiac complications.

Postoperative pain in LC is multifactorial, primarily involving a combination of visceral, referred shoulder, and incisional pain. A multimodal analgesic approach is recommended for pain management. To alleviate LC-related postoperative pain, non-steroidal anti-inflammatory drugs, paracetamol, opioids, local anesthetics, and various regional anesthesia techniques are commonly employed. However, opioids may cause adverse effects, including nausea, vomiting, constipation, and respiratory depression. Neuraxial analgesia is seldom used in LC due to potential complications and technical difficulties. Regional anesthesia and multimodal analgesia have been shown to reduce the neuroendocrine stress response to pain and trauma effectively.

Recently, the use of interfascial plane blocks under ultrasound guidance (USG), considered easy and safe, has increased in LC surgery. The TAP block, first described by Rafi in 2001 and later refined by McDonnell et al. in 2004 as a field block for abdominal surgeries, provides analgesia by blocking the 7th-11th intercostal nerves (T7-T11), the subcostal nerve (T12), and the ilioinguinal (IIN) and iliohypogastric nerves (IHN) (L1-L2). Hebbard et al. later described an ultrasound-guided approach to the TAP block. The recto-intercostal fascial plane block (RIFPB) was introduced in 2023 by Tulgar et al. as an alternative to parasternal intercostal blocks for parasternal surgeries and is reported to block almost the entire upper abdomen. In a case series by Ömür et al., RIFPB was shown to provide both lower sternal and epigastric blockade and sensory block across the upper anterolateral abdomen.

DETAILED DESCRIPTION:
The gallbladder is a small organ located in the upper right quadrant of the abdomen. It stores bile, which helps in the digestion of food. Gallstones are solid bile particles that form due to changes in bile composition and concentration caused by factors such as hormones, medications, diet, and weight changes. Occasionally, a gallstone exits the gallbladder, blocking the normal flow of bile. Acute cholecystitis occurs when the cystic duct is obstructed by a gallstone, causing distension and inflammation of the gallbladder. Cholecystectomy is a commonly performed surgical procedure worldwide for treating acute cholecystitis. Management of acute cholecystitis is divided into medical and surgical approaches. Medical management includes bed rest, analgesic agents, antibiotic therapy, and intravenous fluid replacement. Surgical management involves a procedure called cholecystectomy, the surgical removal of the gallbladder, which can be performed through open or laparoscopic surgery. The laparoscopic technique is superior to open surgery in terms of reduced pain at incision sites, shorter hospital stay, improved quality of life, and faster recovery times. However, although laparoscopic cholecystectomy (LC) is minimally invasive, it can still cause moderate to severe pain. Severe pain can delay postoperative ambulation, reduce patient satisfaction, lead to chronic pain, and increase the risk of pulmonary and cardiac complications.

Postoperative pain in LC has multiple causes. The majority of postoperative pain in LC originates from incision sites (50-70%), pneumoperitoneum (20-30%), and the cholecystectomy procedure itself (10-20%). A multimodal analgesic approach is recommended for pain control. Various analgesic techniques are used to manage postoperative pain caused by LC, including non-steroidal anti-inflammatory drugs, paracetamol, opioids, local anesthetics, and various regional anesthesia techniques. Opioids can lead to side effects such as postoperative nausea and vomiting (PONV), constipation, and respiratory depression. Neuraxial analgesia is rarely used in LC due to potential complications and technical difficulties. The use of regional anesthesia in multimodal analgesia has been shown to significantly reduce the neuroendocrine stress response to pain and trauma.

In recent years, the use of ultrasound-guided (USG) interfascial plane blocks, considered easy and safe, has increased in LC surgeries. The anterolateral abdominal wall consists of the rectus abdominis, external oblique, internal oblique, and transversus abdominis muscles. The transversus abdominis plane, which contains the thoracolumbar nerves from T6-L1, lies between the internal oblique and transversus abdominis muscles. The anterior and lateral abdominal regions are innervated by the anterior branches of the thoracoabdominal nerves from T7-T12 and L1. Therefore, injecting a local anesthetic (LA) into the transversus abdominis plane provides sensory blockade from T7 to L1. TAP block can be part of the analgesic regimen in abdominal surgeries, such as appendectomy, hernia repair, laparotomy, laparoscopic surgeries, cesarean section, abdominal hysterectomy, pyloromyotomy, major abdominal wall surgeries, and colostomy. In another study, Grape et al. reported moderate to high-level evidence that TAP block provided superior analgesia compared to wound infiltration in patients undergoing laparoscopic cholecystectomy.

Tulgar et al. introduced the recto-intercostal fascial plane block (RIFPB) as a novel fascial block for sternotomy and sternal surgeries, reporting that it covers almost the entire upper abdominal region. By injecting LA into the interfascial plane just below the xiphoid process, between the rectus abdominis muscle and the 6th-7th costal cartilages, it blocks the anterior branches. Injection of methylene blue into this plane was observed to spread significantly to the anterior cutaneous branches of the T6-9 nerves and laterally, contributing to abdominal analgesia. Following Tulgar's study, our study aims to target dermatomal coverage between T6-T9 using RIFPB with 20 ml of LA.

Patients will complete the Quality of Recovery-15 (QoR-15) questionnaire, a self-assessment survey that evaluates the quality of postoperative recovery in areas such as physical comfort, pain, independence, psychological support, and emotional state, both on the morning of surgery and 24 hours post-surgery. QoR-15 scores range from 0 to 150, with higher scores indicating better recovery quality. This study will compare the effectiveness of bilateral TAP and bilateral RIFPB in LC, examining postoperative NRS (Numeric Rating Scale) scores, opioid consumption, dermatomal spread, PONV score, and complications to determine which technique is more effective.

ELIGIBILITY:
Inclusion Criteria:

* Will undergo Cholecystectomy surgery
* The American Society of Anesthesiologists (ASA) physical classification is 1-2.
* The volunteer has read and accepted the consent form
* Body mass index (BMI) <35

Exclusion Criteria:

* The patient does not want to participate in the study
* Patients with BMI >35
* Patients with ASA 3-4-5
* Those who are allergic to the local anesthetic used and the specified analgesic drug
* Those who declare that they are during pregnancy and breastfeeding
* Having uncontrollable anxiety
* Those with neuromuscular disease and peripheral nerve diseaseThose who used high doses of opioid medication 3 days before surgery
* Widespread chronic pain, diabetes mellitus, hepatic and renal failure
* Infection at the peripheral block needle insertion site

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-11-10 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Examination with Numeric Rating Scale | 24 hours
  Determination of patients' post-operative pain level. The Numeric Rating Scale (NRS), a method that converts the patient's pain perception into a numerical form, will be used to assess postoperative pain. NRS has a numerical scale ranging from 0 to 10. The patient will rate the intensity of pain on a scale from 0, indicating no pain, to 10, representing the worst imaginable pain (NRS 0=no pain, 4=mild to moderate pain, 6-8=severe pain, and >8=intolerable pain). The NRS score will be evaluated both at rest and during active movement situations (such as transitioning from a lying to a sitting position).

CONTACTS AND LOCATIONS:
Locations (1):
- Hitit University Erol Olcok Training and Research Hospital, Çorum, Turkey (Türkiye)